CLINICAL TRIAL: NCT02192047
Title: Chronic Effects of Natural Palm-based Margarine and Interesterified Palm- and Soy-based Margarine on Insulin Sensitivity and Selected Markers of Cardiovascular Diseases (CVD)
Brief Title: Chronic Effects of Natural and Interesterified Fats Margarine on Insulin Sensitivity and Selected Markers of Cardiovascular Diseases (CVD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malaysia Palm Oil Board (Other Government)
Collaborators: IMU University, Malaysia (Other); Universiti Putra Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PD 174/13
Record Dates: First submitted 2014-06-24; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- palm olein margarine (Experimental): 8 weeks
  Interventions: Other: Palm Olein
- IE palm olein margarine (Experimental): 8 weeks
  Interventions: Other: IE Palm olein
- IE soybean oil-based margarine (Experimental): 8 weeks
  Interventions: Other: IE soybean oil-based

INTERVENTIONS:
Other: Palm Olein — 8 weeks
  Arms: palm olein margarine
Other: IE Palm olein — 8 weeks
  Arms: IE palm olein margarine
Other: IE soybean oil-based — 8 weeks
  Arms: IE soybean oil-based margarine

SUMMARY:
The investigators hypothesized that there will be a significant difference between the effects of trans-free palm-, interesterified palm- and interesterified soybean oil blend on cardiovascular disease, inflammation, insulin resistance and obesity.

DETAILED DESCRIPTION:
Human volunteers will be conditioned for a 8 wk intervention on 3 different test diets providing 30 % energy as fat, 15% energy as protein and 55% energy as carbohydrate according to parallel designed sequences. The test fats used for this study are palm oil, chemically interesterified palm oil and chemically interesterified fully hydrogenated soybean oil and soft oil blend in the form of margarine. Volunteers will be restricted to follow the dietary guidelines throughout the study. Blood collection sessions will held before and after every diet intervention. Outcome measures of the study are serum lipid profile, markers of inflammation, markers of obesity and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females, aged 20-60 yr
* Staff and students of International Medical University, IMU/ Staff of Malaysian Palm Oil Board, MPOB to facilitate centralized consumption of the test fats/snacks
* BMI 21 - 30 kg/m2

Exclusion Criteria:

* Abnomal liver function test (elevated transaminases- alanine aminotransferase,ALT; aspartate aminotransferase,AST))/ abnormal kidney function test (elevated plasma creatinine)
* History of type 2 diabetes mellitus, cancer, stomach ulcers, drug abuse or alcoholism
* Smokers
* On lipid/blood pressure- lowering medication/supplements
* Blood pressure>140/90 mmHg
* Fasting total cholesterol > 6.5 mmol/L
* Fasting TAG > 2.0 mmol/L
* Candidates who are going abroad during the planned schedule for the dietary intervention

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2012-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in serum C-peptide level of subject | up to 8 weeks

SECONDARY OUTCOMES:
Change in serum lipid profile | up to 8 weeks
Change in markers of inflammation | up to 8 weeks
Change in markers of obesity | up to 8 weeks
Change in markers of insulin resistance | up to 8 weeks
Oral Glucose tolerance test (OGTT) | Baseline, month-2

CONTACTS AND LOCATIONS:
Overall Officials: Voon Phooi Tee, Ph.D, Principal Investigator — MPOB; Ng Yen Teng, BSc, Principal Investigator — IMU
Locations (1):
- University Putra Malaysia, Serdang, Selangor, Malaysia